CLINICAL TRIAL: NCT07043114
Title: Influence of Walking Training in Combination With Blood Flow Restriction Training on Muscle Hypertrophy and Quality of Life in PAOD IIa
Brief Title: Impact and Safety of Blood Flow Restriction in Patients With Peripheral Arterial Occlusive Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023_I
Record Dates: First submitted 2025-05-07; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: PAOD (Peripheral Arterial Obstructive Disease)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Patients with PAOD Typ II will perform a six-week walking training with BFR
  Interventions: Other: BFR-Walking

INTERVENTIONS:
Other: BFR-Walking — The training consists of the patients walking on a treadmill twice a week for a total of six weeks until their pain becomes too severe and they have to take a break. After a one-minute break, this is increased again until the pain reaches its maximum. This is done a total of three times per appointment. Additionally, patients will receive a individual BFR intervention bilaterally with a exercise pressure corresponding to 60% of their LOP.

SUMMARY:
In peripheral arterial occlusive disease (PAOD), there is a partial (stenosis) or complete occlusion of peripheral arteries, which leads to reduced arterial blood flow. The cause is atherosclerosis in about 95% of cases and in most cases the lower extremities are affected. The disease is further divided into different stages; stage II is relevant for the present study, specifically IIa. In this case, pain in the legs occurs after a few hundred meters of exertion, e.g. when walking, forcing patients to stop. This condition is also commonly known as intermittent claudication. The therapy of choice is regular gait training, a symptomatic therapy, as the initial cause, atherosclerosis, cannot be treated causally. In the present project, this gait training is supplemented by placing BFR cuffs proximally around the thighs of the patients while walking. The aim is to promote angioneogenesis, which leads to a reduction in symptoms and a corresponding increase in quality of life. A further effect of this can be greater muscle hypertrophy, which also has a positive effect.

DETAILED DESCRIPTION:
Any patient with stage IIa PAOD can be recruited. Patients will complete a walking training with an additionall BFR-pressure applied bilateraly and corresponding to 60% of the individual limb occlusion pressure. The training consists of the patients walking on a treadmill twice a week for a total of six weeks until their pain becomes too severe and they have to take a break. After a one-minute break, this is increased again until the pain reaches its maximum. This is done a total of three times per appointment. After the first three weeks, the intensity of the training is increased by setting a higher speed on the treadmill.

ELIGIBILITY:
Inclusion Criteria:

* PAOD Typ 2
* Eligibitly to exercise on a treadmill

Exclusion Criteria:

* PAOD > Typ 2
* Iatrogenic changes in the vessels of the lower extremities (e.g. Stents)
* Sickle Cell Anemia
* Open Wounds/Infections on the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Pre- (Baseline) to Post-Intervention Phase (after twelve weeks of training intervention)
  Isometric Maximal Strength of the Knee Extensors analyzed by Dynamometer (N)
Quality of Life Score | Pre- (Baseline) to Post-Intervention Phase (after twelve weeks of training intervention)
  Quality of Life assessed by Short-Form 36 Survey

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No